CLINICAL TRIAL: NCT03617380
Title: PharmD Transitions of Care Program (PHARMD-TOC): A Community Pharmacy Transitions of Care Program
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: transferred to different institution
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Candi Morello, Professor Clinical Pharmacy, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 171847
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Disease, Chronic
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHARMD-TOC i (Experimental): PharmD Follow-Up Post Discharge
  Interventions: Other: PharmD TOC
- USUAL CARE (Active Comparator): Usual Post Discharge Procedures
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Usual Care — patients participating Usual Care discharge services
  Arms: USUAL CARE
Other: PharmD TOC — patients participating in a community pharmacy-based Transitions of Care Program (PHARMD-TOC)
  Arms: PHARMD-TOC i

SUMMARY:
Many hospitals and medical groups have developed transitions of care (TOC) programs or procedures in an attempt to reduce hospital readmission and reutilization rates of patients discharged from the hospital. As healthcare's most accessible practitioners, Community Pharmacists have a unique opportunity to assist with reducing unnecessary hospital re-utilization (re-admissions and emergency department visits) after hospital discharge. The purpose of this study is to conduct and evaluate the implementation of a Community Pharmacy-based Transitions of Care (TOC) Program for high-risk post-discharge patients of PIH Health Hospital-Whittier (PIH). The primary objective will be to compare the proportion of patients with hospital re-utilization (readmission, observation status, ED visits) during 30-days post hospital discharge between patients randomly assigned to the PHARMD-TOC group vs. the historic rate at PIH. Secondary analyses will examine differences between groups and describe implementation details of the PHARMD-TOC model of patient care.

ELIGIBILITY:
Inclusion Criteria:

* - Admission LACE Score: in moderate range (5 to 9) And
* Taking high risk medication(s): anticoagulants, insulin, oral antiplatelet agents, oral hypoglycemic agents, opioid analgesics, digoxin Or Taking at least 5 medications AND have one of following: CHF, COPD, Asthma, Pneumonia, Diabetes, ESRD, Schizophrenia, Bi-Polar, Dizziness, History of Falls

And

* Medical or Surgical Unit patients
* Age > 18 years
* Being discharged to home (with or without Home Health services)
* English and/or Spanish speaking
* Will have access to a telephone post-discharge
* Ability to give consent
* Patient admitted to hospital through the emergency department, as a direct admission or as a transfer, or as an elective surgery patient

Exclusion Criteria:

* - Patients with observation status
* Caremore Health Plan patients (Caremore has a separate post-discharge program)
* Patients discharged and followed up by the PIH Coumadin Clinic
* Patients discharged to Residential MD House Calls program
* Patients discharged to Skilled Nursing Facility
* Anyone with planned readmissions
* Obstetrics patients
* Hospice patients
* Oncology patients
* Anyone who does not meet provisions of protocol
* Anyone unwilling or unable to give consent for study procedures and data access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Proportion Patients with Hospital Reutilization | 30 days post hospital discharge
  proportion of patients with hospital re-utilization (readmission, observation status, ED visits) during 30-days post hospital discharge